CLINICAL TRIAL: NCT04627974
Title: A Prospective Study to Evaluate the Long-term Effectiveness, Safety, and Performance of the Saluda Medical's EvokeTM Closed-Loop Spinal Cord Stimulation System to Treat Patients With Chronic Pain of the Trunk and/or Limbs
Brief Title: Long-term Effectiveness, Safety, and Performance of the Evoke Closed-Loop SCS System to Treat Patients With Chronic Pain of the Trunk and/or Limbs
Acronym: Domburg
Status: Active, not recruiting | Type: Observational
Sponsor: Saluda Medical Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-PLC-005299
Record Dates: First submitted 2020-11-06; First posted 2020-11-13 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Spinal Cord Stimulation; Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ECAP-controlled, closed-loop SCS: Spinal cord stimulation that measures and records evoked compound action potentials (ECAPs) and automatically adjusts the stimulation current to maintain a consistent ECAP amplitude
  Interventions: Device: Evoke Spinal Cord Stimulation (SCS) System

INTERVENTIONS:
Device: Evoke Spinal Cord Stimulation (SCS) System — A spinal cord stimulation system that measures and records evoked compound action potentials (ECAPs) and automatically adjusts the stimulation current to maintain a consistent ECAP amplitude

SUMMARY:
The objective of this multicountry, multicentre, prospective study is to evaluate the long-term clinical effectiveness, safety, and performance of the Evoke System in the treatment of chronic pain of the trunk and/or limbs in a real-world population.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for therapy according to the Evoke System indications for use statement and labelling requirements
* Willing and capable of giving informed consent and able to comply with study-related requirements, procedures, and visits
* Baseline VAS pain rating ≥60 mm in the primary area of pain

Exclusion Criteria:

* No further exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic trunk and/or limb pain.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Visual Analogue Scale (VAS) Pain | 3-months post-implant
  Visual Analogue Scale (VAS) to rate pain intensity (0mm [no pain] to 100mm [worst pain imaginable])

SECONDARY OUTCOMES:
Incidence of device- and procedure-related adverse events | through 60-months post-implant
Measurement of ECAPs by the Evoke SCS System | through 60-months post-implant

CONTACTS AND LOCATIONS:
Locations (8):
- Belgium (2):
  - AZ Nikolaas Multidisciplinary Pain Center, Sint-Niklaas, East Flanders
  - AZ Delta Multidisciplinary Pain Center, Roeselare, West Flanders
- Universität Düsseldorf, Düsseldorf, North Rhine-Westphalia, Germany
- Netherlands (2):
  - Erasmus University Medical Center, Rotterdam
  - Rijnstate, Velp
- United Kingdom (3):
  - Basildon University Hospital, Basildon, Essex
  - James Cook University Hospital, Middlesbrough, North Yorkshire
  - Southmead Hospital, Bristol

IPD SHARING:
Plan to Share IPD: No